CLINICAL TRIAL: NCT05719233
Title: Assessment of Neuropsychiatric Function in Patients With Interstitial Lung Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Lecturer of chest diseases and tuberculosis, Assiut University
Other Study IDs: Neuropsychiatric Sequel of ILD
Record Dates: First submitted 2023-01-13; First posted 2023-02-08 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lung Diseases, Interstitial
Keywords: Interstitial lung disease; cognitive function; spirometry; anxiety
MeSH Terms: conditions — Lung Diseases, Interstitial; Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Interstitial Lung disease Group: Mini-mental state examination (MMSE) Hamilton Anxiety Rating Scale Hamilton Depression Rating Scale Nerve conduction studies High resolution Chest Computed tomography Pulmonary function Test
- Control Group: Mini-mental state examination (MMSE) Hamilton Anxiety Rating Scale Hamilton Depression Rating Scale Nerve conduction studies

SUMMARY:
Research on the impact of lung diseases on neuropsychological functioning has revealed impaired cognitive processing in patients with a variety of pulmonary disorders. While the mechanisms responsible for the association of pulmonary diseases and neurocognitive functioning remain unclear, some researchers have attributed it to reduced oxygenation of the brain. Early detection and accurate management of comorbidity have benefits in reducing ILD morbidity and mortality.

DETAILED DESCRIPTION:
Research on the impact of lung diseases on neuropsychological functioning has revealed impaired cognitive processing in patients with a variety of pulmonary disorders. While the mechanisms responsible for the association of pulmonary diseases and neurocognitive functioning remain unclear, some researchers have attributed it to reduced oxygenation of the brain.

Interstitial Lung Disease (ILD) is an "umbrella" term as it comprises a variety of pulmonary diseases which affect the interstitium (the tissue and space around the air sacs of the lungs). It may be caused by a variety of factors (namely, inhaled substances, medications, infection, connective tissue disease, malignancy or idiopathic reasons) and has a clear negative impact on patients' quality of life, leading to symptoms such as fatigue, dyspnea and coughing. Physical sequelae include reduced lung volumes due to tissue thickening, sometimes caused by inflammation. A further consequence is reduced breathing efficiency, resulting in reduced blood oxygen levels and compromised exercise capacity.

Additionally, the fibrosis of the parenchyma impedes the level of gas exchange. A number of studies have reported mood effects in ILD, suggesting, however, that the diagnosis of depression may be obscured, due to the fatigue and apathy that is often a consequence of ILD.

Early detection and accurate management of Neuropsychiatric comorbidities have benefits in reducing ILD morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Interstitial lung disease patients diagnosed using high resolution computed tomography to confirm the diagnosis

Exclusion Criteria:

* Patients who refuse to participate in the study.
* Age less than 18,
* A history of neurological and/or developmental disorders and related drug treatment,
* A head injury with loss of consciousness,
* Active alcohol or drug abuse or a history of abuse prior to testing,
* A history of any psychiatric disorder or treatment, neurological disorders, psychological disorders, dementia, Alzheimer's disease, end-organ failure conditions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Interstitial lung disease patients diagnosed using high resolution computed tomography to confirm the diagnosis either visiting out patient clinic or admitted to ward in assiut university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment | 1 MONTH
  a 30-point test used to assess cognitive function; includes tests of orientation, attention, memory, language, and visual-spatial skills. MMSE score 24-30: no cognitive impairment, 19-23: mild cognitive impairment, 10-18: moderate cognitive impairment, ≤ 9: severe cognitive impairment
Anxiety level | 1 MONTH
  consists of 14 items and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where a score ≤ 17 indicates mild anxiety, 18-24 mild to moderate severity, and more than 24 moderate to severe anxiety
Depression level | 1 MONTH
  The original HAM-D has 21 items, but scoring is based only on the first 17. Scores less than or equal to 7 indicates normal response, 8-13 mild depression, 14-18 Moderate, 19-22 severe, and more than 22 very severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Gamal Elddin Khaleel, Lecturer, Principal Investigator — Assiut university, Egypt
Locations (1):
- Assiut university hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonelli-Incalzi R, Corsonello A, Trojano L, Acanfora D, Spada A, Izzo O, Rengo F. Correlation between cognitive impairment and dependence in hypoxemic COPD. J Clin Exp Neuropsychol. 2008 Feb;30(2):141-50. doi: 10.1080/13803390701287390. PMID 18938666
- [Background] Ryu JH, Daniels CE, Hartman TE, Yi ES. Diagnosis of interstitial lung diseases. Mayo Clin Proc. 2007 Aug;82(8):976-86. doi: 10.4065/82.8.976. PMID 17673067
- [Background] Bors M, Tomic R, Perlman DM, Kim HJ, Whelan TP. Cognitive function in idiopathic pulmonary fibrosis. Chron Respir Dis. 2015 Nov;12(4):365-72. doi: 10.1177/1479972315603552. Epub 2015 Sep 15. PMID 26374298